CLINICAL TRIAL: NCT05742802
Title: A Phase III, Multicentre, Randomised, Double-blind, Chronic-dosing, Parallel-group, Placebo-controlled Extension Study to Evaluate the Long-term Efficacy and Safety of Tozorakimab in Participants With Chronic Obstructive Pulmonary Disease (COPD) With a History of Exacerbations (PROSPERO).
Brief Title: Long-term Efficacy and Safety of Tozorakimab in Participants With Chronic Obstructive Pulmonary Disease With a History of Exacerbations (PROSPERO).
Acronym: PROSPERO
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9180C00008; 2022-501063-41-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2023-01-17; First posted 2023-02-24 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Tozorakimab; MEDI3506; exacerbations; ICS; LABA/LAMA
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tozorakimab Dose 1 (Experimental): Injection subcutaneously Tozorakimab via pre-filled syringe.
  Interventions: Combination Product: Tozorakimab 1
- Tozorakimab Dose 2 (Experimental): Injection subcutaneously Tozorakimab via pre-filled syringe.
  Interventions: Combination Product: Tozorakimab 2
- Placebo (Placebo Comparator): Injection subcutaneously with equivalent volume to Tozorakimab via pre-filled syringe.
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: Tozorakimab 1 — Participants randomised to either dose regimen in the predecessor studies will be assigned to a single Tozorakimab dose regimen in the PROSPERO study.
  Arms: Tozorakimab Dose 1
Combination Product: Tozorakimab 2 — Participants randomised to either dose regimen in the predecessor studies will be assigned to a single Tozorakimab dose regimen in the PROSPERO study.
  Arms: Tozorakimab Dose 2
Combination Product: Placebo — Participants previously randomised to placebo in one of the predecessor studies will be re-randomised in a 1:1 ratio to the active dose of Tozorakimab or placebo.
  Arms: Placebo

SUMMARY:
Subjects who completed either OBERON or TITANIA will be offered the opportunity to consent for this Multicentre, Double-blind, Randomised, Placebo controlled, Parallel Group, Phase 3, extension study to evaluate the safety and efficacy of Tozorakimab in adult participants with symptomatic COPD.

DETAILED DESCRIPTION:
Participants who have completed the study treatment period and have not been prematurely discontinued from IP in one of the predecessor studies, OBERON or TITANIA, will be offered the opportunity to consent for this Multicentre, Double-blind, Randomised, Placebo-controlled, Parallel Group, Phase 3 extension study to evaluate the efficacy and safety of Tozorakimab versus placebo in adult (40 years and older) participants with symptomatic COPD and with a history of exacerbations

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have completed the treatment period and have not been prematurely discontinued from IP in the predecessor studies.
2. Participants who received their last dose of IP in the predecessor studies within the previous 12 weeks and were not withdrawn from the predecessor study.
3. FOCBP (female(s) of childbearing potential) must have a negative urine pregnancy test at Visit 1.
4. Participants who are willing to continue using contraceptive methods as agreed to for the predecessor OBERON or TITANIA studies.
5. Capable of giving signed informed consent.

Exclusion Criteria:

1. Any clinically significant disorder or abnormal findings (clinical, laboratory, instrumental, etc) or major physical and/or cognitive impairment - which, in the opinion of the Investigator, may put the participant at risk because of his/her participation in the study or impact the interpretation of the study results, or otherwise make the participation of the participant inappropriate.
2. Participant meeting criteria for IP discontinuation as judged by the Investigator or the Sponsor.
3. Concurrent enrolment in other interventional clinical studies or treatment with another IP, with the exception of the OBERON and TITANIA predecessor studies.
4. Known history of:

   1. Severe allergic reaction to any monoclonal and polyclonal antibody.
   2. Allergy or reaction to any component of the IP formulation.
5. Chronic use (or expected need for chronic use during the study) of immunosuppressive medications (including, but not limited to, systemic corticosteroids), marketed or investigational biologic, or another prohibited medication.
6. Involvement in the planning and/or conduct of the study (applies to both staff employed by the Sponsor and/or staff at the study site).
7. Participants who are not able to comply with the study requirements, procedures, and restrictions.

Ages: 40 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1711 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2026-02-26 (Estimated); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Annualised rate of severe COPD exacerbations in former smokers. | Up to 104 weeks.
  The primary efficacy endpoint is the rate of severe COPD exacerbations.

SECONDARY OUTCOMES:
The annualised rate of severe COPD exacerbations | Up to 104 weeks.
  To be analyzed as a key secondary endpoint in the Overall Population in former or current smokers.
Time to First Severe COPD Exacerbations | Up to 104 weeks.
  Time to first severe COPD exacerbation over the treatment period. Analyses will be conducted in the former smoker population, followed by the Overall Population in former or current smokers.
Annualised rate of COPD exacerbations requiring hospitalisation and/or ER/ED visits. | Up to 104 weeks.
  To evaluate the long-term effect of Tozorakimab as an add on to SoC compared to with SoC plus placebo on COPD related health care utilisation. Analyses will be conducted in the former smoker population, followed by the Overall Population in former or current smokers.
Time to first moderate-to-severe COPD exacerbation. | Up to 104 weeks.
  To explore the extent to which treatment with each dose of Tozorakimab delays the time to first exacerbation compared with placebo.
Annualised rate of moderate to severe COPD exacerbations. | Up to 104 weeks.
  To evaluate the effect of Tozorakimab as an add on to SoC compared with SoC plus placebo on the rate of moderate to severe COPD exacerbations.
Time to all-cause death. | Up to 104 weeks.
  To evaluate the effect of Tozorakimab as an add on to SoC compared with SoC plus placebo on time to all-cause death.
Trough serum concentrations of Tozorakimab over the treatment period. | Up to 104 weeks.
  Pharmacokinetics: concentrations of Tozorakimab in trough serum.
Incidence of anti-drug antibodies. | Up to 104 weeks.
  Immunogenicity: presence of Tozorakimab anti-drug antibodies in blood serum.

CONTACTS AND LOCATIONS:
Locations (303):
- United States (47):
  - Research Site, Sheffield, Alabama
  - Research Site, Tempe, Arizona
  - Research Site, Lincoln, California
  - Research Site, Newport Beach, California
  - Research Site, Northridge, California
  - Research Site, Boynton Beach, Florida
  - Research Site, Cape Coral, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Plantation, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Evergreen Park, Illinois
  - Research Site, Normal, Illinois
  - Research Site, Greenwood, Indiana
  - Research Site, Kansas City, Kansas
  - Research Site, Bowling Green, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Zachary, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, White Marsh, Maryland
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Toledo, Ohio
  - Research Site, Tulsa, Oklahoma
  - Research Site, DuBois, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Sayre, Pennsylvania
  - Research Site, Rock Hill, South Carolina
  - Research Site, Franklin, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Boerne, Texas
  - Research Site, Kingwood, Texas
  - Research Site, McKinney, Texas
  - Research Site, Tomball, Texas
  - Research Site, Colchester, Vermont
  - Research Site, Williamsburg, Virginia
  - Research Site, Cudahy, Wisconsin
- Argentina (10):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, Quilmes
  - Research Site, San Fernando
  - Research Site, San Juan Bautista
  - Research Site, San Miguel de Tucumán
- Australia (9):
  - Research Site, Campbelltown
  - Research Site, Frankstown
  - Research Site, Macquarie University
  - Research Site, Melbourne
  - Research Site, Nedlands
  - Research Site, Southport
  - Research Site, Spearwood
  - Research Site, Wollongong
  - Research Site, Woodville South
- Belgium (5):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Namur
- Brazil (8):
  - Research Site, Blumenau
  - Research Site, Botucatu
  - Research Site, Brasília
  - Research Site, Curitiba
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São Bernardo do Campo
  - Research Site, São Paulo
- Bulgaria (9):
  - Research Site, Dupnitsa
  - Research Site, Kozloduy
  - Research Site, Lovech
  - Research Site, Petrich
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Sliven
  - Research Site, Sofia
  - Research Site, Vratsa
- Canada (7):
  - Research Site, Edmonton, Alberta
  - Research Site, Sherwood Park, Alberta
  - Research Site, Ajax, Ontario
  - Research Site, Guelph, Ontario
  - Research Site, Winchester, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Chile (4):
  - Research Site, Chile
  - Research Site, Curicó
  - Research Site, Santiago
  - Research Site, Talca
- China (29):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Hohhot
  - Research Site, Kunming
  - Research Site, Linhai
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xiamen
  - Research Site, Xuzhou
  - Research Site, Yangzhou
  - Research Site, Yinchuan
  - Research Site, Zhanjiang
  - Research Site, Zunyi
- Colombia (4):
  - Research Site, Barranquilla
  - Research Site, Ibagué
  - Research Site, Rionegro
  - Research Site, Zipaquirá
- Czechia (5):
  - Research Site, Brno
  - Research Site, Jindřichův Hradec
  - Research Site, Liberec
  - Research Site, Olomouc
  - Research Site, Rokycany
- Denmark (6):
  - Research Site, Aalborg
  - Research Site, Copenhagen
  - Research Site, Hvidovre
  - Research Site, Næstved
  - Research Site, Roskilde
  - Research Site, Vejle
- Finland (4):
  - Research Site, Hämeenlinna
  - Research Site, Helsinki
  - Research Site, Kuopio
  - Research Site, Turku
- France (9):
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Dijon
  - Research Site, La Tronche
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Toulouse
- Germany (8):
  - Research Site, Ahrensburg
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Darmstadt
  - Research Site, Halle
  - Research Site, Marburg
  - Research Site, Peine
- Greece (6):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Exohi Thessaloniki
  - Research Site, Ioannina
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Hungary (7):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Edelény
  - Research Site, Encs
  - Research Site, Mosonmagyaróvár
  - Research Site, Nyíregyháza-Sóstóhegy
  - Research Site, Százhalombatta
- India (8):
  - Research Site, Belagavi
  - Research Site, Coimbatore
  - Research Site, Dehradun
  - Research Site, Jaipur
  - Research Site, Nagpur
  - Research Site, Nashik
  - Research Site, New Delhi
  - Research Site, Thane
- Israel (6):
  - Research Site, Ashkelon
  - Research Site, Beersheba
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Rehovot
  - Research Site, Tel Aviv
- Italy (12):
  - Research Site, Bari
  - Research Site, Carrara
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Roma
  - Research Site, Salerno
  - Research Site, Sassari
  - Research Site, Statte
  - Research Site, Telese Terme
  - Research Site, Tradate
  - Research Site, Vercelli
  - Research Site, Verona
- Japan (22):
  - Research Site, Asahikawa-shi
  - Research Site, Fujieda-shi
  - Research Site, Fukuoka
  - Research Site, Hamamatsu
  - Research Site, Hiroshima
  - Research Site, Iizuka-shi
  - Research Site, Itabashi-ku
  - Research Site, Iwata-shi
  - Research Site, Kanazawa
  - Research Site, Kawachinagano-shi
  - Research Site, Kobe
  - Research Site, Matsusaka-shi
  - Research Site, Mizunami-shi
  - Research Site, Nagoya
  - Research Site, Obihiro
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Shinjuku-ku
  - Research Site, Shizuoka
  - Research Site, Toshima-ku
  - Research Site, Toyonaka-shi
  - Research Site, Yokohama
- Mexico (8):
  - Research Site, Benito Juárez
  - Research Site, Chihuahua City
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Morelia
  - Research Site, Oaxaca City
  - Research Site, Veracruz
- Netherlands (5):
  - Research Site, Eindhoven
  - Research Site, Groningen
  - Research Site, Harderwijk
  - Research Site, Heerlen
  - Research Site, Zutphen
- Norway (3):
  - Research Site, Lørenskog
  - Research Site, Oslo
  - Research Site, Tønsberg
- Research Site, Lima, Peru
- Philippines (3):
  - Research Site, Baguio City
  - Research Site, Cebu City
  - Research Site, Iloilo City
- Poland (11):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Ostrowiec Świętokrzyski
  - Research Site, Ostróda
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Sosnowiec
  - Research Site, Wroclaw
- Portugal (4):
  - Research Site, Guimarães
  - Research Site, Lisbon
  - Research Site, Matosinhos Municipality
  - Research Site, Vila Franca de Xira
- Romania (4):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Timișoara
- South Korea (4):
  - Research Site, Daegu
  - Research Site, Incheon
  - Research Site, Jeonju
  - Research Site, Seoul
- Spain (8):
  - Research Site, Galdakao
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Mérida
  - Research Site, Pozuelo de Alarcón
  - Research Site, Santander
  - Research Site, Valencia
  - Research Site, Zaragoza
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Lund
  - Research Site, Stockholm
- Taiwan (6):
  - Research Site, Hsinchu
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
  - Research Site, Yunlin
- Thailand (7):
  - Research Site, Bang Kra So
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Muang,
  - Research Site, Muang
  - Research Site, Mueang
  - Research Site, Nakhon Ratchasima
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Mersin
- United Kingdom (6):
  - Research Site, Bradford
  - Research Site, Corby
  - Research Site, High Wycombe
  - Research Site, Northwood
  - Research Site, Preston
  - Research Site, Shipley
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home